CLINICAL TRIAL: NCT01135667
Title: Thrombocytes And IndividuaLization of ORal Antiplatelet Treatment After Percutaneous Coronary Intervention
Brief Title: Prasugrel Versus Double Dose Clopidogrel to Treat Clopidogrel Low-responsiveness After PCI
Acronym: TAILOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lene Holmvang (Other)
Responsible Party: Sponsor-Investigator, Lene Holmvang, MD DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAILOR
Record Dates: First submitted 2010-04-23; First posted 2010-06-03 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Acute Coronary Syndromes
Keywords: clopidogrel; prasugrel; low responder; multiplate; verify now
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clopidogrel (Active Comparator): clopidogrel 150 mg once daily for 30 days (and then 75 mg for additional 11 months - not study related)
  Interventions: Drug: clopidogrel
- Prasugrel (Active Comparator): Prasugrel 10 mg once daily for 30 days (and then clopidogrel 75 mg once daily for additional 11 months - not study related)
  Interventions: Drug: Prasugrel 10 mg

INTERVENTIONS:
Drug: clopidogrel — clopidogrel 150 mg once daily for 30 days
  Other Names: Plavix
  Arms: clopidogrel
Drug: Prasugrel 10 mg — Prasugrel 10 mg once daily for 30 days
  Other Names: Efient
  Arms: Prasugrel

SUMMARY:
All patients undergoing elective or sub-acute PCI are screened by MULTIPLATE test for clopidogrel low-responsiveness after receiving 600 mg clopidogrel the day before.

A cut off value has previously been established. Only low-responders with Multiplate values above the cut off value are included in the study. The patients are randomized to either clopidogrel 150 mg once daily or Prasugrel 10 mg (age > 75 og bodyweight < 60 kg 5 mg)once daily for 30 days after the procedure.

Follow up will be at 30 days after PCI were another MULTIPLATE test will be performed.

Primary endpoint:Platelet inhibition (by MULTIPLATE) after 30 days of intensified antiplatelet therapy.

Clinical endpoints such as bleeding complications (GUSTO, TIMI) during treatment, and major adverse cardiac events (MACE) at 30 days will be collected and reported but the study size does not allow for formal statistical analysis The study ends by the 30 days follow up visit and all patients continue with clopidogrel 75 mg once daily for another 11 months (not study related)

ELIGIBILITY:
Inclusion Criteria:

* PCI with stenting and Multiplate hep-ADP > 70 U despite clopidogrel loading

Exclusion Criteria:

* need for vit K antagonist
* women with childbearing potential
* breastfeeding women
* Planned surgery within 6 months
* Intolerance to clopidogrel, prasugrel or aspirin
* previous stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Heparin ADP by Multiplate | 30 days
  Test of platelet inhibition (ADP receptor mediated) after 30 days of intensifiet anti platelet therapy

CONTACTS AND LOCATIONS:
Overall Officials: Lene Holmvang, MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Department of Cardiology, 2013, Copenhagen O, Denmark